CLINICAL TRIAL: NCT06180967
Title: A Phase I, Open Label, Fixed-sequence Drug Interaction Study to Investigate the Effect of Multiple Oral Doses of LOXO-305 on the Pharmacokinetics of a Single Dose of Intravenous and Oral Midazolam (CYP3A4 Substrate) in Healthy Subjects
Brief Title: A Drug Drug Interaction (DDI) Study of Pirtobrutinib (LOXO-305) and Different Formulations of Midazolam in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Loxo Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: LOXO-BTK-20008; J2N-OX-JZND (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — pirtobrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Midazolam (Intravenous [IV] Bolus) (Experimental): A single IV bolus dose of midazolam will be administered in the morning following a 10-hour fast prior to dosing and a 4-hour fast postdose on Day 1 and Day 15.
  Interventions: Drug: Midazolam Solution
- Midazolam Oral (Experimental): A single oral dose of midazolam will be administered in the morning following a 10-hour fast prior to dosing and a 4-hour fast postdose on Day 3 and Day 17.
  Interventions: Drug: Midazolam Syrup
- Pirtobrutinib (Experimental): Multiple oral doses of Pirtobrutinib once a day (QD) will be administered on Days 5 through Day 17.
  Interventions: Drug: Pirtobrutinib

INTERVENTIONS:
Drug: Midazolam Syrup — Administered Orally.
  Arms: Midazolam Oral
Drug: Midazolam Solution — Administered IV bolus.
  Arms: Midazolam (Intravenous [IV] Bolus)
Drug: Pirtobrutinib — Administered Orally.
  Other Names: LOXO-305; LY3527727
  Arms: Pirtobrutinib

SUMMARY:
The main purpose of this study is to assess the effect of Pirtobrutinib (LOXO-305) on how fast different formulations of midazolam gets into the blood stream and how long it takes the body to remove it when administered in healthy participants. The study will also access how much endogenous coproporphyrins I and III as biomarkers of OATP1B1 and OATP1B3 is in the bloodstream and how the body handles and eliminates them following single and multiple oral doses of Pirtobrutinib. Safety and tolerability of Pirtobrutinib will also be evaluated. For each participant, the total duration of the study will be 59 days, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Must have Body mass index (BMI) within the range of 18.0 to 32.0 kilograms per square meter (kg/m²), inclusive
* Male and female participants in good health, determined by no clinically significant findings from medical history, 12-lead Electrocardiogram (ECG), vital sign measurements, or clinical laboratory evaluations as assessed by the investigator
* Female participants of non-childbearing potential and male participants who follow standard contraceptive methods
* Must have comply with all study procedures, including the 8-night stay at the Clinical Research Unit (CRU) and follow-up phone call

Exclusion Criteria:

* History or presence of any diseases or conditions of clinical significance by the Investigator (or designee) and/or Sponsor
* Positive serologic test for hepatitis B surface antigen (HBsAg), hepatitis B virus immunoglobulin M (HBV IgM) core antibody, hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antibody at Screening
* Positive polymerase chain reaction (PCR) test for COVID-19 at Screening or Check-in (Day -1)
* Known ongoing alcohol and/or drug abuse within 2 years prior to Screening
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee)
* Have previously completed or withdrawn from any other study investigating Pirtobrutinib (LOXO-305) and have previously received the investigational product

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renee Ward, MD, PhD, Study Director — Loxo Oncology, Inc.
Locations (1):
- Covance Clinical Research Unit, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of 2 periods: Period 1 and Period 2. A total of 15 healthy participants were enrolled in the study.
Groups:
- Period 1: All Participants: Midazolam (IV + Oral Dose): * Day 1: Participants received a single intravenous (IV) bolus dose of midazolam 250 micrograms (mcg) solution on Day 1.
  * Day 3: Participants received a single oral dose of midazolam 500 mcg syrup on Day 3.
  A washout period of 2 days between midazolam IV dose and midazolam oral dose on Day 1 and Day 3 was observed.
- Period 2: All Participants: Pirtobrutinib + Midazolam (IV + Oral Dose): * Day 5-17: Participants received Pirtobrutinib 200 mg tablets orally once daily (QD) in the morning from Day 5 through Day 17;
  * Day 15: Participants received single IV bolus dose of Midazolam 250 mcg followed by Pirtobrutinib intake on Day 15.
  * Day 17: Participants received a single oral dose of midazolam 500 mcg syrup followed by Pirtobrutinib intake on Day 17.
  A washout period of 2 days between midazolam IV dose and midazolam oral dose on Day 15 and Day 17 was observed.
Period: Period 1: Day 1 to Day 4
Arm/Group | Period 1: All Participants: Midazolam (IV + Oral Dose) | Period 2: All Participants: Pirtobrutinib + Midazolam (IV + Oral Dose)
Started | 15 | 0
Received at Least 1 Dose of Study Drug | 15 | 0
Completed | 15 | 0
Not Completed | 0 | 0
Period: Period 2: Day 5 to Day 20
Arm/Group | Period 1: All Participants: Midazolam (IV + Oral Dose) | Period 2: All Participants: Pirtobrutinib + Midazolam (IV + Oral Dose)
Started | 0 | 15 (Participants who completed Period 1 continued to receive treatment in Period 2.)
Received at Least 1 Dose of Study Drug | 0 | 15
Completed | 0 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- All Participants: Midazolam (IV + Oral Dose) + Pirtobrutinib: All participants in the study who received:
  * Period 1, Day 1: Participants received a single intravenous (IV) bolus dose of midazolam 250 micrograms (mcg) solution on Day 1.
  * Period 1 Day 3: Participants received a single oral dose of midazolam 500 mcg syrup on Day 3. A washout period of 2 days between midazolam IV dose and midazolam oral dose on Day 1 and Day 3 was observed.
  * Period 2, Day 5-17: Participants received Pirtobrutinib 200 mg tablets orally once daily (QD) in the morning from Day 5 through Day 17
  * Period 2, Day 15: Participants received single IV bolus dose of Midazolam 250 mcg followed by Pirtobrutinib intake on Day 15.
  * Period 2, Day 17: Participants received a single oral dose of midazolam 500 mcg syrup followed by Pirtobrutinib intake on Day 17. A washout period of 2 days between midazolam IV dose and midazolam oral dose on Day 15 and Day 17 was observed.
Arm/Group | All Participants: Midazolam (IV + Oral Dose) + Pirtobrutinib
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (9.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 10
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration-Time Curve From Hour 0 to the Last Measurable Concentration (AUC0-t) of Midazolam and Its Metabolite 1-hydroxymidazolam (1-OH-midazolam) Following Oral Dose Administration
Description: PK: AUC0-t of midazolam and its metabolite 1-OH-midazolam following oral dose administration was reported.
Time Frame: Period 1: Day 3 (pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post-dose); Period 2: Day 17 (pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post-dose)
Population: All participants who received at least 1 dose of oral midazolam had at least 1 quantifiable PK concentration, and for whom at least 1 PK parameter was computed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms per milliliter (h*ng/mL)
Groups:
- Period 1: Oral Midazolam 500 mcg (Day 3): Participants who received a single oral dose of midazolam 500 mcg syrup on Day 3.
- Period 2: Pirtobrutinib 200 mg + Oral Midazolam 500 mcg (Day 17): Participants who received pirtobrutinib 200 mg tablets orally followed by a single oral dose of midazolam 500 mcg syrup on Day 17.
Arm/Group | Period 1: Oral Midazolam 500 mcg (Day 3) | Period 2: Pirtobrutinib 200 mg + Oral Midazolam 500 mcg (Day 17)
Number analyzed (Participants) | 15 | 15
Hours*nanograms per milliliter (h*ng/mL)
  Midazolam | 4.81 (40.8) | 8.30 (43.2)
  Metabolite: 1-OH-medazolam | 2.24 (41.9) | 2.52 (40.6)

2. Primary Outcome: PK: Area Under the Concentration-Time From Time 0 Extrapolated To Infinity (AUC0-inf) of Midazolam and Its Metabolite 1-OH-Midazolam Following Oral Dose Administration
Description: PK: AUC(0-inf) of midazolam and its metabolite 1-OH-midazolam following oral dose administration was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1: Oral Midazolam 500 mcg (Day 3) | Period 2: Pirtobrutinib 200 mg + Oral Midazolam 500 mcg (Day 17)
Number analyzed (Participants) | 15 | 15
h*ng/mL
  Midazolam | 5.31 (43.1) | 9.01 (44.0)
  Metabolite: 1-OH-midazolam | 2.60 (39.9) | 2.92 (42.2)

3. Primary Outcome: PK: Percentage Extrapolation for AUC0-inf (%AUCextrap) of Midazolam and Its Metabolite 1-OH-Midazolam Following Oral Dose Administration
Description: PK: %AUCextrap of midazolam and its metabolite 1-OH-midazolam following oral dose administration was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUC0-inf
Arm/Group | Period 1: Oral Midazolam 500 mcg (Day 3) | Period 2: Pirtobrutinib 200 mg + Oral Midazolam 500 mcg (Day 17)
Number analyzed (Participants) | 15 | 15
percentage of AUC0-inf
  Midazolam | 8.84 (33.7) | 7.42 (35.3)
  Metabolite: 1-OH-midazolam | 12.9 (37.5) | 12.2 (48.6)

4. Primary Outcome: PK: Maximum Observed Plasma Concentration (Cmax) of Midazolam and Its Metabolite 1-OH-Midazolam Following Oral Dose Administration
Description: PK: Cmax of midazolam and its metabolite 1-OH-midazolam following oral dose administration was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Period 1: Oral Midazolam 500 mcg (Day 3) | Period 2: Pirtobrutinib 200 mg + Oral Midazolam 500 mcg (Day 17)
Number analyzed (Participants) | 15 | 15
nanograms per milliliter (ng/mL)
  Midazolam | 2.33 (36.7) | 3.68 (34.3)
  Metabolite: 1-OH-midazolam | 1.25 (42.2) | 1.41 (40.2)

5. Primary Outcome: PK: Time to Maximum Observed Plasma Concentration (Tmax) of Midazolam and Its Metabolite 1-OH-Midazolam Following Oral Dose Administration
Description: PK: tmax of midazolam and its metabolite 1-OH-midazolam following oral dose administration was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Period 1: Oral Midazolam 500 mcg (Day 3) | Period 2: Pirtobrutinib 200 mg + Oral Midazolam 500 mcg (Day 17)
Number analyzed (Participants) | 15 | 15
Hours
  Midazolam | 0.750 [0.500 to 1.00] | 0.500 [0.500 to 0.750]
  Metabolite: 1-OH-midazolam | 0.750 [0.500 to 1.00] | 0.500 [0.500 to 1.00]

6. Primary Outcome: PK: Apparent Terminal Elimination Rate Constant (Lambda [λ] z) of Midazolam and Its Metabolite 1-OH-Midazolam Following Oral Dose Administration
Description: PK: λz of midazolam and its metabolite 1-OH-midazolam following oral dose administration was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: one per hour (1/h)
Arm/Group | Period 1: Oral Midazolam 500 mcg (Day 3) | Period 2: Pirtobrutinib 200 mg + Oral Midazolam 500 mcg (Day 17)
Number analyzed (Participants) | 15 | 15
one per hour (1/h)
  Midazolam | 0.316 (50.7) | 0.227 (50.2)
  Metabolite: 1-OH-midazolam | 0.441 (35.4) | 0.419 (61.2)

7. Primary Outcome: PK: Apparent Systemic Clearance (CL/F) of Midazolam Following Oral Dose Administration
Description: PK: CL/F of midazolam following oral dose administration was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour (L/h)
Arm/Group | Period 1: Oral Midazolam 500 mcg (Day 3) | Period 2: Pirtobrutinib 200 mg + Oral Midazolam 500 mcg (Day 17)
Number analyzed (Participants) | 15 | 15
Liters per hour (L/h) | 94.2 (43.1) | 55.5 (44.0)

8. Primary Outcome: PK: Apparent Volume of Distribution (Vz/F) of Midazolam Following Oral Dose Administration
Description: PK: Vz/F of midazolam following oral dose administration was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Period 1: Oral Midazolam 500 mcg (Day 3) | Period 2: Pirtobrutinib 200 mg + Oral Midazolam 500 mcg (Day 17)
Number analyzed (Participants) | 15 | 15
Liters | 298 (29.7) | 244 (29.6)

9. Primary Outcome: PK: Apparent Plasma Terminal Elimination Half-life (t½) of Midazolam and Its Metabolite 1-OH-Midazolam Following Oral Dose Administration
Description: PK: t½ of midazolam and its metabolite 1-OH-midazolam following oral dose administration was reported.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Period 1: Oral Midazolam 500 mcg (Day 3) | Period 2: Pirtobrutinib 200 mg + Oral Midazolam 500 mcg (Day 17)
Number analyzed (Participants) | 15 | 15
hours
  Midazolam | 2.20 (50.7) | 3.05 (50.2)
  Metabolite: 1-OH-midazolam | 1.57 (35.4) | 1.65 (61.2)

10. Primary Outcome: PK: Total Clearance (CL) of Midazolam Following Intravenous Dose Administration
Description: PK: CL of midazolam following intravenous dose administration was reported.
Time Frame: Period 1: Day 1 (pre-dose, 5 minutes, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post-dose); Period 2: Day 15 (pre-dose, 5 minutes, 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours post-dose)
Population: All participants who received at least 1 dose of IV midazolam had at least 1 quantifiable PK concentration, and for whom at least 1 PK parameter was computed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Groups:
- Period 1: IV Midazolam 250 mcg (Day 1): Participants who received a single IV bolus dose of midazolam 250 mcg solution on Day 1.
- Period 2: Pirtobrutinib 200 mg + IV Midazolam 250 mcg (Day 15): Participants who received pirtobrutinib 200 mg tablets orally followed by IV bolus dose of midazolam 250 mcg solution on Day 15.
Arm/Group | Period 1: IV Midazolam 250 mcg (Day 1) | Period 2: Pirtobrutinib 200 mg + IV Midazolam 250 mcg (Day 15)
Number analyzed (Participants) | 15 | 15
L/h | 26.0 (21.4) | 23.1 (26.5)

11. Primary Outcome: PK: Volume of Distribution (Vz) of Midazolam Following Intravenous Dose Administration
Description: PK: Vz of midazolam following intravenous dose administration was reported.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Period 1: IV Midazolam 250 mcg (Day 1) | Period 2: Pirtobrutinib 200 mg + IV Midazolam 250 mcg (Day 15)
Number analyzed (Participants) | 15 | 15
Liters | 113 (34.2) | 105 (37.8)

12. Primary Outcome: PK: Volume of Distribution at Steady State (Vss) of Midazolam Following Intravenous Dose Administration
Description: PK: Vss of midazolam following intravenous dose administration was reported.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Period 1: IV Midazolam 250 mcg (Day 1) | Period 2: Pirtobrutinib 200 mg + IV Midazolam 250 mcg (Day 15)
Number analyzed (Participants) | 15 | 15
Liters | 78.2 (29.4) | 76.1 (31.0)

13. Primary Outcome: PK: Area Under the Concentration-Time Curve From Hour 0 to the Last Measurable Concentration (AUC0-t) of Midazolam and Its Metabolite 1-OH-midazolam Following Intravenous Dose Administration
Description: PK: AUC0-t of midazolam and its metabolite 1-OH-midazolam following intravenous dose administration was reported.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1: IV Midazolam 250 mcg (Day 1) | Period 2: Pirtobrutinib 200 mg + IV Midazolam 250 mcg (Day 15)
Number analyzed (Participants) | 15 | 15
h*ng/mL
  Midazolam | 8.89 (21.6) | 10.1 (25.1)
  Metabolite: 1-OH-medazolam | 1.39 (41.7) | 1.21 (35.7)

14. Primary Outcome: PK: Area Under the Concentration-Time From Time 0 Extrapolated To Infinity (AUC0-inf) of Midazolam and Its Metabolite 1-OH-midazolam Following Intravenous Dose Administration
Description: PK: AUC0-inf of midazolam and its metabolite 1-OH-midazolam following intravenous dose administration was reported.
Time Frame: as for outcome 10
Population: All participants who received at least 1 dose of IV midazolam had at least 1 quantifiable PK concentration, and for whom at least 1 PK parameter was computed. Here, 'Number analyzed' signifies participants with available data for each specified category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 1: IV Midazolam 250 mcg (Day 1) | Period 2: Pirtobrutinib 200 mg + IV Midazolam 250 mcg (Day 15)
Number analyzed (Participants) | 15 | 15
h*ng/mL
  Midazolam | 9.62 (21.4) | 10.8 (26.5)
  Metabolite: 1-OH-medazolam: number analyzed (Participants) | 7 | 8
  Metabolite: 1-OH-medazolam | 2.13 (43.0) | 1.62 (25.2)

15. Primary Outcome: PK: Percentage Extrapolation for AUC0-inf (%AUCextrap) of Midazolam and Its Metabolite 1-OH-midazolam Following Intravenous Dose Administration
Description: PK: %AUCextrap of midazolam and its metabolite 1-OH-midazolam following intravenous dose administration was reported.
Time Frame: as for outcome 10
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUC0-inf
Arm/Group | Period 1: IV Midazolam 250 mcg (Day 1) | Period 2: Pirtobrutinib 200 mg + IV Midazolam 250 mcg (Day 15)
Number analyzed (Participants) | 15 | 15
percentage of AUC0-inf
  Midazolam | 7.13 (37.1) | 6.44 (42.0)
  Metabolite: 1-OH-medazolam: number analyzed (Participants) | 7 | 8
  Metabolite: 1-OH-medazolam | 19.6 (24.7) | 24.7 (11.5)

16. Primary Outcome: PK: Maximum Observed Plasma Concentration (Cmax) of Midazolam and Its Metabolite 1-OH-midazolam Following Intravenous Dose Administration
Description: PK: Cmax of midazolam and its metabolite 1-OH-midazolam following intravenous dose administration was reported.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Period 1: IV Midazolam 250 mcg (Day 1) | Period 2: Pirtobrutinib 200 mg + IV Midazolam 250 mcg (Day 15)
Number analyzed (Participants) | 15 | 15
ng/mL
  Midazolam | 6.96 (34.8) | 6.91 (27.8)
  Metabolite: 1-OH-medazolam | 0.512 (31.7) | 0.475 (28.6)

17. Primary Outcome: PK: Time to Maximum Observed Plasma Concentration (Tmax) of Midazolam and Its Metabolite 1-OH-midazolam Following Intravenous Dose Administration
Description: PK: tmax of midazolam and its metabolite 1-OH-midazolam following intravenous dose administration was reported.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Median (Full Range); unit: hours
Arm/Group | Period 1: IV Midazolam 250 mcg (Day 1) | Period 2: Pirtobrutinib 200 mg + IV Midazolam 250 mcg (Day 15)
Number analyzed (Participants) | 15 | 15
hours
  Midazolam | 0.0833 [0.0833 to 0.250] | 0.0833 [0.0833 to 0.0833]
  Metabolite: 1-OH-medazolam | 0.750 [0.500 to 1.00] | 0.750 [0.500 to 1.00]

18. Primary Outcome: PK: Apparent Terminal Elimination Rate Constant (λz) of Midazolam and Its Metabolite 1-OH-midazolam Following Intravenous Dose Administration
Description: PK: λz of midazolam and its metabolite 1-OH-midazolam following intravenous dose administration was reported.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Period 1: IV Midazolam 250 mcg (Day 1) | Period 2: Pirtobrutinib 200 mg + IV Midazolam 250 mcg (Day 15)
Number analyzed (Participants) | 15 | 15
1/h
  Midazolam | 0.229 (37.0) | 0.221 (49.5)
  Metabolite: 1-OH-medazolam | 0.224 (55.7) | 0.282 (47.8)

19. Primary Outcome: PK: Apparent Plasma Terminal Elimination Half-life (t½) of Midazolam and Its Metabolite 1-OH-midazolam Following Intravenous Dose Administration
Description: PK: t1/2 of midazolam and its metabolite 1-OH-midazolam following intravenous dose administration was reported.
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Period 1: IV Midazolam 250 mcg (Day 1) | Period 2: Pirtobrutinib 200 mg + IV Midazolam 250 mcg (Day 15)
Number analyzed (Participants) | 15 | 15
hours
  Midazolam | 3.02 (37.0) | 3.13 (49.5)
  Metabolite: 1-OH-medazolam | 3.09 (55.7) | 2.46 (47.8)

20. Secondary Outcome: PK: Area Under the Concentration-Time Curve From Hour 0 to the Last Measurable Concentration (AUC0-t) of Pirtobrutinib
Description: PK: AUC0-t of Pirtobrutinib was reported.
Time Frame: Period 2: Day 5, Day 14 and Day 15 (pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24 hours post-dose), Day 17 (pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, and 100 hours post-dose)
Population: The PK population included all participants who received at least 1 dose of pirtobrutinib had at least 1 quantifiable PK concentration, and for whom at least 1 PK parameter was computed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Period 2: Pirtobrutinib 200 mg (Day 5): Participants who received pirtobrutinib 200 mg tablets orally on Day 5.
- Period 2: Pirtobrutinib 200 mg (Day 14): Participants who received pirtobrutinib 200 mg tablets orally on Day 14.
- Period 2: Pirtobrutinib 200 mg + Oral Midazolam 500 mcg (Day 17): Participants who received pirtobrutinib 200 mg tablets orally followed by oral dose of midazolam 500 mcg syrup on Day 17.
Arm/Group | Period 2: Pirtobrutinib 200 mg (Day 5) | Period 2: Pirtobrutinib 200 mg (Day 14) | Period 2: Pirtobrutinib 200 mg + IV Midazolam 250 mcg (Day 15) | Period 2: Pirtobrutinib 200 mg + Oral Midazolam 500 mcg (Day 17)
Number analyzed (Participants) | 15 | 15 | 15 | 15
h*ng/mL | 54800 (20.0) | 114000 (26.0) | 115000 (25.0) | 211000 (33.8)

21. Secondary Outcome: PK: Area Under the Concentration-time Curve During a Dosing Interval (AUCtau) of Pirtobrutinib
Description: PK: AUCtau of Pirtobrutinib was reported.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Period 2: Pirtobrutinib 200 mg (Day 5) | Period 2: Pirtobrutinib 200 mg (Day 14) | Period 2: Pirtobrutinib 200 mg + IV Midazolam 250 mcg (Day 15) | Period 2: Pirtobrutinib 200 mg + Oral Midazolam 500 mcg (Day 17)
Number analyzed (Participants) | 15 | 15 | 15 | 15
h*ng/mL | 55000 (20.0) | 114000 (26.1) | 116000 (25.0) | 118000 (25.5)

22. Secondary Outcome: PK: Maximum Observed Plasma Concentration (Cmax) of Pirtobrutinib
Description: PK: Cmax of Pirtobrutinib was reported.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Period 2: Pirtobrutinib 200 mg + Oral Midazolam 500 mcg (Day 17): Participants who received pirtobrutinib 200 mg tablets orally in followed by oral dose of midazolam 500 mcg syrup on Day 17.
Arm/Group | Period 2: Pirtobrutinib 200 mg (Day 5) | Period 2: Pirtobrutinib 200 mg (Day 14) | Period 2: Pirtobrutinib 200 mg + IV Midazolam 250 mcg (Day 15) | Period 2: Pirtobrutinib 200 mg + Oral Midazolam 500 mcg (Day 17)
Number analyzed (Participants) | 15 | 15 | 15 | 15
ng/mL | 4880 (18.5) | 8120 (27.1) | 8620 (23.1) | 8750 (27.2)

23. Secondary Outcome: PK: Concentration Observed at the End Of the Dosing Interval (Ctrough) of Pirtobrutinib
Description: PK: Ctrough of Pirtobrutinib before multiple oral doses administration was reported.
Time Frame: Period 2: 24-hour post-dose on Day 14, Day 15, and Day 17
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Period 2: Pirtobrutinib 200 mg (Day 14) | Period 2: Pirtobrutinib 200 mg + IV Midazolam 250 mcg (Day 15) | Period 2: Pirtobrutinib 200 mg + Oral Midazolam 500 mcg (Day 17)
Number analyzed (Participants) | 15 | 15 | 15
ng/mL | 3060 (32.1) | 3180 (36.4) | 3050 (32.7)

24. Secondary Outcome: PK: Time To Maximum Observed Plasma Concentration (Tmax) of Pirtobrutinib
Description: PK: tmax of Pirtobrutinib was reported.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Median (Full Range); unit: hours
Arm/Group | Period 2: Pirtobrutinib 200 mg (Day 5) | Period 2: Pirtobrutinib 200 mg (Day 14) | Period 2: Pirtobrutinib 200 mg + IV Midazolam 250 mcg (Day 15) | Period 2: Pirtobrutinib 200 mg + Oral Midazolam 500 mcg (Day 17)
Number analyzed (Participants) | 15 | 15 | 15 | 15
hours | 2.50 [1.00 to 4.00] | 3.00 [2.00 to 4.00] | 3.00 [0.750 to 6.00] | 3.00 [1.00 to 4.00]

25. Secondary Outcome: PK: Apparent Systemic Plasma Clearance at Steady State (CL,ss/F) of Pirtobrutinib
Description: PK: CL,ss/F of Pirtobrutinib was reported.
Time Frame: Period 2: Day 14 and Day 15 (pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24 hours post-dose), Day 17 (pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 48, 72, and 100 hours post-dose)
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Period 2: Pirtobrutinib 200 mg (Day 14) | Period 2: Pirtobrutinib 200 mg + IV Midazolam 250 mcg (Day 15) | Period 2: Pirtobrutinib 200 mg + Oral Midazolam 500 mcg (Day 17)
Number analyzed (Participants) | 15 | 15 | 15
L/h | 1.75 (26.1) | 1.72 (25.0) | 1.69 (25.5)

26. Secondary Outcome: PK: Accumulation Ratio (RAUC) of Pirtobrutinib
Description: RAUC was ratio of Day 14 AUCtau to Day 5 AUCtau.
Time Frame: Period 2: Day 5 and Day 14 (pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, and 24 hours post-dose)
Population: as for outcome 20
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Groups:
- Period 2: Pirtobrutinib 200 mg: Participants received Pirtobrutinib 200 mg tablets orally once daily (QD) in the morning from Day 5 through Day 17.
Arm/Group | Period 2: Pirtobrutinib 200 mg
Number analyzed (Participants) | 15
Ratio | 2.08 (15.9)

ADVERSE EVENTS:
Time Frame: From Day 1 up to 7 days post end of treatment (i.e., up to Day 30)
Description: All participants who received at least 1 dose of study drugs (pirtobrutinib, IV midazolam, or oral midazolam). Participants were classified into groups based on actual treatment received.
Groups:
- Period 1: IV Midazolam 250 mcg: Participants received a single IV bolus dose of midazolam 250 mcg solution on Day 1.
- Period 1: Oral Midazolam 500 mcg: Participants received a single oral dose of midazolam 500 mcg syrup on Day 3
- Period 2: Pirtobrutinib 200 mg: Participants received pirtobrutinib 200 mg tablets orally QD from Day 5 through Day 17.
- Period 2: Pirtobrutinib 200 mg + IV Midazolam 250 mcg: Participants received pirtobrutinib 200 mg tablets orally followed by IV bolus dose of midazolam 250 mcg solution on Day 15.
- Period 2: Pirtobrutinib 200 mg + Oral Midazolam 500 mcg: Participants received pirtobrutinib 200 mg tablets orally followed by oral dose of midazolam 500 mcg syrup on Day 17.
Arm/Group | Period 1: IV Midazolam 250 mcg | Period 1: Oral Midazolam 500 mcg | Period 2: Pirtobrutinib 200 mg | Period 2: Pirtobrutinib 200 mg + IV Midazolam 250 mcg | Period 2: Pirtobrutinib 200 mg + Oral Midazolam 500 mcg
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/15 | 0/15 | 3/15 | 1/15 | 0/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: IV Midazolam 250 mcg (N=15) | Period 1: Oral Midazolam 500 mcg (N=15) | Period 2: Pirtobrutinib 200 mg (N=15) | Period 2: Pirtobrutinib 200 mg + IV Midazolam 250 mcg (N=15) | Period 2: Pirtobrutinib 200 mg + Oral Midazolam 500 mcg (N=15)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-09-13): https://cdn.clinicaltrials.gov/large-docs/67/NCT06180967/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-16): https://cdn.clinicaltrials.gov/large-docs/67/NCT06180967/SAP_001.pdf